CLINICAL TRIAL: NCT04419675
Title: The Course of Low Back Pain: a Prospective Cohort Study
Brief Title: The Course of Low Back Pain
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 109643
Record Dates: First submitted 2020-05-27; First posted 2020-06-05 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2021-10

CONDITIONS: Low Back Pain; Type of Leg Pain (Radicular, Non-radicular); Lifestyle (Sedentary Behavior and Physical Activity); Start Back Screening Tool
MeSH Terms: conditions — Low Back Pain; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational Cohort, usual care = physical therapy — usual care = physical therapy

SUMMARY:
This study aims to research the possible associations of education level, sedentary lifestyle, and type of low back pain (radicular vs non-radicular) with the course of low back pain and recovery rate.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain
* Age 18 years or older

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with low back pain contacting physical therapy for treatment of low back pain
Sampling Method: Non-Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Functional Limitations | Measurement at baseline
  Measured with Patient Specific Scale (0=no limitation, 100=impossible to perform) and Oswestry Disability Index (0=no limitation, 100=very limited)
Functional Limitations | Measurement at 6 weeks
  Measured with Patient Specific Scale (0=no limitation, 100=impossible to perform) and Oswestry Disability Index (0=no limitation, 100=very limited)
Functional Limitations | Measurement at 12 weeks
  Measured with Patient Specific Scale (0=no limitation, 100=impossible to perform) and Oswestry Disability Index (0=no limitation, 100=very limited)
Functional Limitations | Measurement at 26 weeks
  Measured with Patient Specific Scale (0=no limitation, 100=impossible to perform) and Oswestry Disability Index (0=no limitation, 100=very limited)
Functional Limitations | Measurement at 52 weeks
  Measured with Patient Specific Scale (0=no limitation, 100=impossible to perform) and Oswestry Disability Index (0=no limitation, 100=very limited)
Recovery rate | 26 weeks after inclusion
  Global Perceived Effect (7-point Likert-scale where 0=much worse, 7=completely recovered)
Recovery rate | 52 weeks after inclusion
  Global Perceived Effect (7-point Likert-scale where 0=much worse, 7=completely recovered)
Pain with Numeric Pain Rating Scale | measurement at baseline
  Numeric Pain Rating Scale (0= no pain, 10= maximum pain)
Pain with Numeric Pain Rating Scale | measurement at 6 weeks
  Numeric Pain Rating Scale (0= no pain, 10= maximum pain)
Pain with Numeric Pain Rating Scale | measurement at 12 weeks
  Numeric Pain Rating Scale (0= no pain, 10= maximum pain)
Pain with Numeric Pain Rating Scale | measurement at 26 weeks
  Numeric Pain Rating Scale (0= no pain, 10= maximum pain)
Pain with Numeric Pain Rating Scale | measurement at 52 weeks
  Numeric Pain Rating Scale (0= no pain, 10= maximum pain)

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (6):
  - Fysius Amersfoort, Amersfoort
  - Fysius Arnhem, Arnhem
  - Fysius Eindhoven, Eindhoven
  - Fysius Nijmegen, Nijmegen
  - Fysius Rotterdam, Rotterdam
  - Fysius Winterswijk, Winterswijk

IPD SHARING:
Plan to Share IPD: Undecided
Storage at central data storage of Radboud University Medical Center